CLINICAL TRIAL: NCT04543357
Title: A Low-Interventional Study Of AAV9 Neutralizing Antibody Seroconversion in Household Contacts of Participants Within the C3391003 Clinical Trial
Brief Title: A Study to Evaluate AAV9 Neutralizing Antibody Seroconversion in Household Contacts.
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to lack of efficacy in the Phase 3 study C3391003, Pfizer has decided to terminate any future dosing of fordadistrogene movaparvovec.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3391007; ARISEN (Other: Alias Study Number)
Record Dates: First submitted 2020-08-07; First posted 2020-09-10 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Household Contacts
Keywords: seroconversion; viral shedding; DNA vector shedding
MeSH Terms: conditions — HIV Seropositivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Household contacts of a DMD patient in an interventional study of fordadistrogene movaparvovec.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood Samples for NAb and ADA to AAV9

SUMMARY:
This study will include male and female participants who live or work in the same household as a patient in one of the fordadistrogene movaparvovec interventional studies. Up to 5 participants from the same household may be enrolled. The objective is to estimate the likelihood of NAb seroconversion to AAV9 in household contacts of a patient in one of the interventional studies who is treated with fordadistrogene movaparvovec gene therapy.

DETAILED DESCRIPTION:
This single center study will include approximately 50 to 250 participants and is designed to estimate the likelihood of NAb seroconversion to AAV9 because of exposure to shed viral vector material released by a DMD patient treated with fordadistrogene movaparvovec in an interventional study. Eligible participants will undergo a blood draw provided by a Home Health Care Vendor at three home visits.

The total duration of participation in this study is about 4 months, including up to 48 days for the screening/baseline period and about 56 days after the DMD patient of the same household is dosed with the investigational gene therapy in the interventional study.

To maintain the blind in the blinded interventional studies, all C3391007 study participants and investigators as well as the sponsor will remain blinded to the Cohort assignment of the interventional study patient until the interventional study becomes unblinded.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who weigh at least 9 kg.
* Anticipated to be living or working in the same household as a patient in one of the fordadistrogene movaparvovec interventional studies for at least 4 months.
* Anticipated to have > 10 hours of contact per week and expected to have direct contact with the interventional study patient.
* The interventional patient is dosed in the interventional study.

Exclusion Criteria:

* Prior treatment with gene therapy utilizing AAV vectors of any serotype.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This single center study will include approximately 50 to 250 participants who live or work in the same household as a DMD patient in one of the fordadistrogene movaparvovec interventional studies. Up to 5 participants from the same household may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a low-interventional study to assess development of neutralizing Antibodies (NAbs) to adeno associated virus serotype 9 (AAV9) in household contacts of Duchenne Muscular Dystrophy (DMD) Patients Treated with fordadistrogene movaparvovec.
Groups:
- Participants With Potential Fordadistrogene Movaparvovec Exposure: People working or living in the same household of patients who were enrolled in an interventional study of fordadistrogene movaparvovec (including study C3391003 [NCT04281485] and C3391002 [not listed on ClinicalTrials.gov]) were enrolled.
Period: Overall Study
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who signed the informed consent document, and 1) who were household members of interventional study participants (including siblings) who were assigned to fordadistrogene movaparvovec or placebo and received a single dose of study treatment and 2) who had at least one day of contact with the interventional study participant during the first 2 weeks.
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Previously Seronegative for Neutralizing Antibodies [NAbs] to AAV9) Who Developed NAb to AAV9 at Day 28 After the Interventional Study Patient Was Dosed
Description: Development of NAb to AAV9 was defined by an increase of >=6-fold above Baseline titer in participants with a detectable, but negative test (ie, titer >=1 and <4) for NAb to AAV9 at Baseline. If there was an undetectable titer at Baseline (ie, titer <1), then development of NAb to AAV9 was defined by a NAb to AAV9 titer >=6.
Time Frame: Day 28 after the interventional study participant was dosed
Population: "Number of participants analyzed" signifies number of participants evaluable for the outcome measure: Participants with a NAb titer undetectable (ie, titer <1) or detectable, but negative test (ie, titer >=1 and <4) at Baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Participants (Previously Seronegative for Anti-Drug Antibody [ADA] to AAV9) Who Developed ADA to AAV9 at Day 28 After the Interventional Study Patient Was Dosed
Description: Development of ADA to AAV9 was defined by a titer ≥300 in participants with a negative test (ie, titer <50) for ADA to AAV9 at Baseline.
Time Frame: Day 28 after the interventional study participant was dosed
Population: "Number of participants analyzed" signifies number of participants evaluable for the outcome measure: Participants with an ADA titer negative at Baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Number analyzed (Participants) | 7
Participants | 0

3. Primary Outcome: Number of Participants (Previously Seronegative for NAb to AAV9) Who Developed NAb to AAV9 at Day 56 After the Interventional Study Patient Was Dosed
Description: as for outcome 1
Time Frame: Day 56 after the interventional study participant was dosed
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Number of Participants (Previously Seronegative for Anti-Drug Antibody [ADA] to AAV9) Who Developed ADA to AAV9 at Day 56 After the Interventional Study Patient Was Dosed
Description: as for outcome 2
Time Frame: Day 56 after the interventional study participant was dosed
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from Screening (Day -48 to Day -1) up to Day 56.
Description: MedDRA v26
Arm/Group | Participants With Potential Fordadistrogene Movaparvovec Exposure
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04543357/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT04543357/SAP_001.pdf